CLINICAL TRIAL: NCT02768701
Title: Phase II Study Of Single-dose Cyclophosphamide +Pembrolizumab In Patients With Metastatic Triple Negative Breast Cancer
Brief Title: Study Of Single-dose Cyclophosphamide +Pembrolizumab In Patients With Metastatic Triple Negative Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCCC 1525
Record Dates: First submitted 2016-05-05; First posted 2016-05-11 (Estimated); Results first posted 2022-08-03 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-05

CONDITIONS: Triple Negative Breast Cancer
Keywords: Pembrolizumab; cyclophosphamide
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — pembrolizumab; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Experimental: Single Arm (Experimental): Subjects will receive a single dose (300 mg/m2) of cyclophosphamide given the day before cycle 1 of pembrolizumab (200 mg), which will be administered every 3 weeks.
  Interventions: Drug: Pembrolizumab; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Pembrolizumab — Subjects will be treated every 3 weeks with 200 mg of pembrolizumab via a 30 minute infusion.
  Other Names: Keytruda
Drug: Cyclophosphamide — A single 300 mg/m2 dose of cyclophosphamide IV over 30-60 minutes will be administered on Day 1 of this study.
  Other Names: Cytoxan; Neosar

SUMMARY:
The purpose of this study is to evaluate pembrolizumab therapy in patients with triple-negative breast cancer (TNBC) who have received at least one prior line of therapy.

DETAILED DESCRIPTION:
This phase II, single-arm, multicenter study will evaluate efficacy and toxicity of administration of pembrolizumab following cyclophosphamide therapy, in advanced stage triple-negative breast cancer.

Duration of Therapy

Treatment may continue until one of the following occurs:

* Disease progression
* Inter-current illness that prevents further administration of treatment
* Unacceptable adverse event(s)
* Pregnancy
* Patient decides to withdraw from study treatment,
* General or specific changes in the patient's condition render the patient unacceptable for further treatment in the judgment of the investigator
* Completed 24 months of uninterrupted treatment with pembrolizumab or 35 administrations of study medication, whichever is later

Duration of Follow Up

* Subjects will be followed for up to 3 years after removal from study treatment or until death, whichever occurs first.
* Patients removed from study for unacceptable adverse events (AEs) will be followed until resolution or stabilization of the event(s).

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent and HIPAA authorization for release of personal health information. NOTE: HIPAA authorization may be included in the informed consent or obtained separately.
2. Age ≥ 18 years at the time of consent.
3. Have measurable disease based on RECIST 1.1 (see section 6.7 for details).
4. ECOG Performance Status ≤ 1 as defined in the protocol ECOG Performance Status.
5. Subject must have histologically confirmed stage IV TNBC (ER-, PR-, HER2-negative) and have received at least 1 prior line of systemic therapy.

   * ER- and PR-negative: defined as < 1% staining by immunohistochemistry (IHC)
   * HER2-negative disease, defined as IHC 0-1+ or fluorescence in situ hybridization (FISH) ratio < 2.0
6. Patients with stable brain metastases will be allowed provided the following criteria are met:

   * Brain radiation was already provided at least 4 weeks prior to initiating study treatment
   * The subject has no new or progressive neurologic symptoms AND neurological symptom stability for the last 4 weeks prior to the study
   * The subject has been off of corticosteroids for at least 7 days prior to trial treatment
   * The subject does not have carcinomatous meningitis
7. Demonstrate adequate organ function as defined in the table below; all screening labs to be obtained within 72 h of initiating study treatment.
8. Females of childbearing potential must have a negative serum pregnancy test within 72 hrs prior to treatment. NOTE: Females are considered of child bearing potential unless they are surgically sterile, have a congenital acquired condition that prevents childbearing (have undergone a hysterectomy, bilateral tubal ligation/occlusion, bilateral salpingectomy or bilateral oophorectomy at least 6 weeks prior to screening) or they are naturally postmenopausal for at least 12 consecutive months without an alternative medical cause. In women < 45 years of age a high follicle stimulating hormone level in the postmenopausal range may be used to confirm a post-menopausal state in women not using hormonal contraception or hormonal replacement therapy. In the absence of 12 months of amenorrhea, a single FSH measurement is insufficient.
9. Female patients of childbearing potential should be willing to use appropriate birth control as outlined in Section 5.2.8, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication.
10. Male subjects of childbearing potential must agree to use an adequate method of contraception as outlined in Section 5.2.8, starting with the first dose of study therapy through 120 days after the last dose of study therapy.
11. Consent for the use of any residual material from biopsy (archival tissue) and serial blood draws will be required for enrollment; fresh biopsy (pre and post dose) of tumor tissue will be optional. NOTE: Patients without adequate tissue for bio correlates will not be excluded or required to have a repeat biopsy.
12. As determined by the enrolling physician or protocol designee, the subject should be able to understand and comply with study procedures for the entire length of the study.
13. Has a LVEF within the normal institutional range (or ≥ 50%) based on ECHO or MUGA.

Exclusion Criteria:

1. Active infection requiring systemic therapy
2. Pregnant or breastfeeding (NOTE: breast milk cannot be stored for future use while the mother is being treated on study).
3. Has a known history of active Bacillus Tuberculosis (TB)
4. Hypersensitivity to pembrolizumab or any of its excipients.
5. Has a known additional malignancy that is active and/or progressive requiring treatment; exceptions include basal cell or squamous cell skin cancer, in situ cervical or bladder cancer, or other cancer for which the subject has been disease-free for at least five years.
6. Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to receipt of study medication or who has not recovered (i.e., ≤ Grade 1 or at baseline; excludes alopecia and Grade 2 neuropathy) from adverse events due to a previously administered agent.

   • If subject had major surgery, they must have recovered adequately from the toxicity and complications from the intervention prior to starting therapy
7. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
8. Has had monoclonal antibody therapy within 4 weeks prior to study Day 1 or who has not recovered (ie, ≤ Grade 1 at baseline; excludes alopecia and Grade 2 neuropathy) from adverse events due to agent(s) administered more than 4 weeks earlier.
9. Treatment with any investigational drug within 4 weeks or 5 half-lives, whichever is shorter, prior to the first dose of study medication.
10. Used an investigational device within 4 weeks of the first dose of treatment.
11. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
12. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg, thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
13. Has known history of, or any evidence of active, non-infectious pneumonitis requiring treatment with steroids; has history of, or any evidence of, active interstitial lung disease.
14. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
15. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
16. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
17. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
18. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
19. Has participated in a previous trial and received pembrolizumab therapy
20. Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
21. Has received a live vaccine within 30 days prior to the first dose of trial treatment.

    • Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed
22. Cyclophosphamide is a substrate for cytochromes 2B6, 2C9, 3A4 and 2C19. Patients must not have received any drug that is a moderate or strong inhibitor of 2B6, 2C9, 3A4, and 2C19 within 1 week prior to receiving cyclophosphamide dosing through 72 hours after cyclophosphamide dosing. Patients must not have received any drug that is a moderate or strong inducer of 3A4 within 2 weeks prior to cyclophosphamide dosing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-10-18 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2023-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth C Dees, MD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (5):
- United States (5):
  - George Washington University-Medical Faculty Associates, Washington D.C., District of Columbia
  - Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Cone Health Cancer Center, Greensboro, North Carolina
  - Rex Cancer Center, Raleigh, North Carolina
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: UNC Lineberger Comprehensive Cancer Center — http://unclineberger.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled at five institutions (UNC-Chapel Hill, University of Pittsburgh, Moses Cone, UNC-Rex Cancer Center, and George Washington University) from November, 2016 to February, 2018. All subjects started to receive study treatment in November 2016 although 2 subjects signed informed consent in October 2016.
Pre-assignment Details: A total of forty-nine subjects consented to the study, but eight were deemed to be ineligible and one subject has withdrawn the consent during screening. Forty subjects were enrolled and evaluable for toxicity and survival, and 39 subjects were evaluable for response.
Period: Overall Study
Arm/Group | Experimental: Single Arm
Started | 40
Completed | 32
Not Completed | 8

BASELINE CHARACTERISTICS:
Arm/Group | Experimental: Single Arm
Number analyzed (Participants) | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 32
  >=65 years | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 28
  More than one race | 1
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 40
ECOG performance status [Count of Participants; unit: Participants] — East Coast Oncology Group (ECOG) Performance status : 0-5 scale to describe a patient's level of functioning in terms of selfcare ability and activity level (lower score means higher functioning) 0-Fully active
  1-Restricted in strenuous activity but ambulatory and able to carry out light work
  Participants
    0 | 24
    1 | 16
Stage at diagnosis [Count of Participants; unit: Participants] — American Cancer Society Clinical Staging system that considers tumor size, tumor spread to lymph nodes and other parts of the body, and tumor cell characteristics used. Stage 0 is non-invasive carcinoma, and stages I through IV are invasive breast cancer, stage IV is tumor spreads to other parts of the body. Increasing stages result in worse treatment outcomes.
  Participants
    0-III | 30
    IV | 10
Prior (neo)adjuvant therapy [Count of Participants; unit: Participants]
  Yes | 33
  No | 7
Sites of metastatic disease [Count of Participants; unit: Participants]
  Liver | 12
  Lung | 14
  Bone | 18
  Lymph node | 4
  Brain | 1

OUTCOME MEASURES:

1. Primary Outcome: The Progression Free Survival (PFS)
Description: PFS is defined as the time from day1 of the study treatment until disease progression or death. Disease progression is defined as per Response Evaluation Criteria In Solid Tumors Criteria (RECIST)1.1 based on computerized tomography (CT), magnetic resonance imaging (MRI), or positron emission tomography (PET) images or assessment of the physician.
  RECIST v.1.1: Complete Response (CR), disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Stable Disease (SD), no response or less response than Partial or Progressive; or Progressive Disease (PD), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: Up to 5 years
Population: The subjects received at least one dose of the study treatment were included.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Experimental: Single Arm
Number analyzed (Participants) | 35
months | 1.8 [1.4 to 2.3]

2. Primary Outcome: Quantification of the Change in Regulatory T Cells (Tregs) During the Study Treatment.
Description: Regulatory T cells (Tregs) are counted before the treatment start and during the treatment. Methods: Blood Sample collection.
Time Frame: Up to 2 years
Population: The subjects received two doses of the study treatment.
Measure: Median (Full Range); unit: Percent Change in Tregs
Groups:
- C1D1-C1D2: Changes in Tregs count value from Cycle 1 Day 1 to Cycle 1 Day 2
- C1D1-C2D1: Changes in Tregs count value from Cycle 1 Day 1 to Cycle 2 Day 1
- C1D2-C2D1: Changes in Tregs count value from Cycle 1 Day 2 to Cycle 2 Day 1
Arm/Group | C1D1-C1D2 | C1D1-C2D1 | C1D2-C2D1
Number analyzed (Participants) | 40 | 40 | 40
Percent Change in Tregs | -3.3 [-67.1 to 258.3] | 10 [-62 to 143.5] | 21.7 [-54 to 169.9]

3. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR is defined as the percentage of patients with [compete response (CR) + partial response (PR)] per RECIST1.1 based on computerized tomography (CT), magnetic resonance imaging (MRI), or positron emission tomography (PET) images.
  RECIST v.1.1: Complete Response (CR), disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions;
Time Frame: Up to 2 years
Population: The subjects received at least one dose of the study treatment and treatments response was assessed.
Measure: Number; unit: percentage of participants
Arm/Group | Experimental: Single Arm
Number analyzed (Participants) | 39
percentage of participants | 21

4. Secondary Outcome: Duration of Response (DOR)
Description: DOR is defined as the time from documentation of tumor response by RECIST1.1 [(CR) + (PR)] to disease progression by RECIST 1.1. It will be measured from when the time measurement criteria are first met for complete response or partial response (whichever status is recorded first) until the first date of progressive disease or death. Patients who neither progress nor die will be censored on the date of their last tumor assessment.
Time Frame: Up to 3 years
Population: The subjects received at least one dose of the study treatment and treatments response was assessed.
Measure: Median (Full Range); unit: months
Arm/Group | Experimental: Single Arm
Number analyzed (Participants) | 39
months | 20.4 [2 to 34]

5. Secondary Outcome: Disease Control Rate (DCR)
Description: DCR is defined as the percentage of participants, who achieve [compete response (CR) + partial response (PR) and stable disease (SD) per RECIST1.1. If best response is SD, then it must last more than 6 months to be included in calculation of DCR, to be considered to have received clinical benefit from the treatment regimen.
  RECIST v.1.1: Complete Response (CR), disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Stable Disease (SD), no response or less response than Partial or Progressive; or Progressive Disease (PD), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: Up to 2 years
Population: The subjects received the study treatment, treatments response was assessed and/or followed up for more than 6 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental: Single Arm
Number analyzed (Participants) | 39
Participants | 28

6. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from D1 of study treatment to death from any cause.
Time Frame: Up to 3 years
Population: All subjects who received at least one dose of treatment were included.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Experimental: Single Arm
Number analyzed (Participants) | 35
months | 6.3 [2.8 to 9.3]

7. Secondary Outcome: Treatment Associated Toxicity
Description: Treatment Associated Toxicity is defined as the number of participants with Grade 3-4 adverse events associated with study treatment.
  Adverse Events were classified and graded according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v.4 based on changes in laboratory parameters, vital signs, and other safety assessments per standard of care.
Time Frame: Up to 3 years
Population: Participants who received at least one cycle of study treatment were included.
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental: Single Arm
Number analyzed (Participants) | 40
Participants
  White blood cell decreased | 2
  Pericardial tamponade | 1
  Pain | 1
  Neutrophil count decreased | 2
  Lymphocyte count decreased | 1
  Immune system disorders | 1
  Hypoalbuminemia | 1
  Headache | 1
  Generalized muscle weakness | 1
  Gastrointestinal disorders | 1
  Fatigue | 3
  Dyspnea | 2
  Dry mouth | 1
  Diarrhea | 2
  Colitis | 1
  Blood bilirubin increased | 1
  Aspartate aminotransferase increased | 2
  Anorexia | 1
  Anemia | 2
  Alkaline phosphatase increased | 1
  Alanine aminotransferase increased | 1

ADVERSE EVENTS:
Time Frame: From day 1 of the study treatment up to 3 years
Description: Treatment Associated Toxicity will be graded number of participants with Adverse Events. Adverse Events will be classified and graded according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) criteria v4.0 based on changes in laboratory parameters, vital signs, and other safety assessments per standard of care.
Arm/Group | Experimental: Single Arm
All-Cause Mortality (participants affected / at risk) | 5/40
Serious Adverse Events (participants affected / at risk) | 18/40
Other Adverse Events (participants affected / at risk) | 40/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental: Single Arm (N=40)
Anemia (Blood and lymphatic system disorders) | 1
Pericardial tamponade (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Supraventricular tachycardia (Cardiac disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Colitis (Gastrointestinal disorders) | 1
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1
Colonic perforation (Gastrointestinal disorders) | 1
Pain (General disorders) | 1
Fever (General disorders) | 1
Infections and infestations - Other, specify (Infections and infestations) | 1
Sepsis (Infections and infestations) | 2
Investigations - Other, specify (Investigations) | 1
Alkaline phosphatase increased (Investigations) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Lethargy (Nervous system disorders) | 1
Presyncope (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 1
Nervous system disorders - Other, specify (Nervous system disorders) | 1
Paresthesia (Nervous system disorders) | 1
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental: Single Arm (N=40)
Anemia (Blood and lymphatic system disorders) | 28
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 1
Leukocytosis (Blood and lymphatic system disorders) | 1
Lymph node pain (Blood and lymphatic system disorders) | 5
Cardiac disorders - Other, specify (Cardiac disorders) | 3
Palpitations (Cardiac disorders) | 2
Pericardial effusion (Cardiac disorders) | 1
Pericardial tamponade (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 6
Supraventricular tachycardia (Cardiac disorders) | 1
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 1
Hearing impaired (Ear and labyrinth disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Vertigo (Ear and labyrinth disorders) | 3
Endocrine disorders - Other, specify (Endocrine disorders) | 2
Hyperthyroidism (Endocrine disorders) | 5
Hypothyroidism (Endocrine disorders) | 9
Blurred vision (Eye disorders) | 1
Dry eye (Eye disorders) | 4
Eye disorders - Other, specify (Eye disorders) | 3
Scleral disorder (Eye disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 8
Ascites (Gastrointestinal disorders) | 1
Bloating (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 21
Diarrhea (Gastrointestinal disorders) | 12
Dry mouth (Gastrointestinal disorders) | 5
Dyspepsia (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 2
Gastroesophageal reflux disease (Gastrointestinal disorders) | 9
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 2
Mucositis oral (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 20
Oral dysesthesia (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 7
Chills (General disorders) | 3
Edema face (General disorders) | 2
Edema limbs (General disorders) | 13
Fatigue (General disorders) | 30
Fever (General disorders) | 2
Flu like symptoms (General disorders) | 1
General disorders and administration site conditions - Other, specify (General disorders) | 7
Irritability (General disorders) | 2
Non-cardiac chest pain (General disorders) | 2
Pain (General disorders) | 11
Immune system disorders - Other, specify (Immune system disorders) | 1
Infections and infestations - Other, specify (Infections and infestations) | 4
Lung infection (Infections and infestations) | 1
Mucosal infection (Infections and infestations) | 2
Rash pustular (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Upper respiratory infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 5
Bruising (Injury, poisoning and procedural complications) | 1
Fracture (Injury, poisoning and procedural complications) | 2
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 2
Spinal fracture (Injury, poisoning and procedural complications) | 2
Activated partial thromboplastin time prolonged (Injury, poisoning and procedural complications) | 2
Alanine aminotransferase increased (Investigations) | 12
Alkaline phosphatase increased (Investigations) | 8
Aspartate aminotransferase increased (Investigations) | 17
Blood bilirubin increased (Investigations) | 3
Cholesterol high (Investigations) | 3
Creatinine increased (Investigations) | 4
Investigations - Other, specify (Investigations) | 2
Lymphocyte count decreased (Investigations) | 25
Neutrophil count decreased (Investigations) | 7
Platelet count decreased (Investigations) | 2
Weight gain (Investigations) | 1
Weight loss (Investigations) | 3
White blood cell decreased (Investigations) | 11
Acidosis (Metabolism and nutrition disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 13
Dehydration (Metabolism and nutrition disorders) | 1
Glucose intolerance (Metabolism and nutrition disorders) | 1
Hypercalcemia (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 5
Hyperkalemia (Metabolism and nutrition disorders) | 2
Hypernatremia (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 15
Hypocalcemia (Metabolism and nutrition disorders) | 7
Hypoglycemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 9
Hypomagnesemia (Metabolism and nutrition disorders) | 10
Hyponatremia (Metabolism and nutrition disorders) | 15
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 6
Arthritis (Musculoskeletal and connective tissue disorders) | 4
Back pain (Musculoskeletal and connective tissue disorders) | 8
Bone pain (Musculoskeletal and connective tissue disorders) | 4
Chest wall pain (Musculoskeletal and connective tissue disorders) | 4
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 3
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 5
Myositis (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 4
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8
Akathisia (Nervous system disorders) | 1
Amnesia (Nervous system disorders) | 1
Brachial plexopathy (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 4
Dysarthria (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 2
Headache (Nervous system disorders) | 9
Memory impairment (Nervous system disorders) | 1
Nervous system disorders - Other, specify (Nervous system disorders) | 1
Neuralgia (Nervous system disorders) | 1
Paresthesia (Nervous system disorders) | 2
Peripheral motor neuropathy (Nervous system disorders) | 2
Peripheral sensory neuropathy (Nervous system disorders) | 17
Presyncope (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 1
Sinus pain (Nervous system disorders) | 2
Somnolence (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Agitation (Psychiatric disorders) | 2
Anxiety (Psychiatric disorders) | 17
Confusion (Psychiatric disorders) | 2
Depression (Psychiatric disorders) | 9
Insomnia (Psychiatric disorders) | 17
Libido decreased (Psychiatric disorders) | 2
Restlessness (Psychiatric disorders) | 1
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 3
Urinary frequency (Renal and urinary disorders) | 3
Urinary incontinence (Renal and urinary disorders) | 3
Urinary urgency (Renal and urinary disorders) | 3
Urine discoloration (Renal and urinary disorders) | 1
Breast pain (Reproductive system and breast disorders) | 2
Pelvic pain (Reproductive system and breast disorders) | 1
Reproductive system and breast disorders - Other, specify (Reproductive system and breast disorders) | 1
Vaginal dryness (Reproductive system and breast disorders) | 3
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 15
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 17
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 8
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 3
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 3
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 6
Body odor (Skin and subcutaneous tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 4
Pain of skin (Skin and subcutaneous tissue disorders) | 2
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 4
Rash acneiform (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 7
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 10
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
Surgical and medical procedures - Other, specify (Skin and subcutaneous tissue disorders) | 1
Flushing (Vascular disorders) | 1
Hematoma (Vascular disorders) | 1
Hot flashes (Vascular disorders) | 5
Hypertension (Vascular disorders) | 16
Lymphedema (Vascular disorders) | 11
Thromboembolic event (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-22): https://cdn.clinicaltrials.gov/large-docs/01/NCT02768701/Prot_SAP_000.pdf